CLINICAL TRIAL: NCT04461067
Title: Ultrasonographic Evaluation of the Evolution of the Gastric Volume After Colorectal
Brief Title: Gastric Volume and Colorectal Surgery
Acronym: EVOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19.12.02.56807
Record Dates: First submitted 2020-06-24; First posted 2020-07-08 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2021-07

CONDITIONS: Postoperative Ileus
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gastric antrum measurement (Experimental)
  Interventions: Diagnostic Test: ultrasonography

INTERVENTIONS:
Diagnostic Test: ultrasonography — Ultrasonography of the stomach is performed to measure the diameter of the antrum

SUMMARY:
Postoperative ileus (POI) is a serious complication after colorectal surgery. One of its most frequent consequences is the replacement of nasogastric tube because of the vomiting. Vomiting is due to the distension of the stomach and information on the evolution of gastric filling after surgery could help to better understand the physiopathology of POI. It could also give indication to help the physician in the management of POI.

The ultrasonography has been shown to be a reliable technic to assess the gastric emptying.

To date, there is no indication in the literature about the evolution of the gastric filling after colorectal surgery while these information could help to identify patients at risk for POI and to predict the need for POI replacement.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing colorectal resection whatever the surgical access

Exclusion Criteria:

* contra-indication to ultrasonography performance
* history of gastrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-08 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Diameter of the gastric antrum | immediately before the procedure and each postoperative day up to discharge (mean 7 days)

SECONDARY OUTCOMES:
postoperative ileus | in the morning up to 30 postoperative days
Postoperative quality of life: GIQLI | before discharge
  GIQLI
postoperative morbidity | within 30 postoperative days
  Dindo Clavien Scale (from 1 (minor) to 5 (death))

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien VENARA, MD, PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Venara A, Paisant A, Gillet J, Morgado L, Rebmann E, Hamel JF. The ultrasonographic measure of postoperative day 2 gastric volume may be a useful tool to improve the management of colorectal surgery patients: results of an ancillary study. Int J Colorectal Dis. 2026 Jan 27;41(1):48. doi: 10.1007/s00384-026-05092-z. PMID 41588201